CLINICAL TRIAL: NCT04292405
Title: Accuracy of Cardiac Acoustic Biomarkers Recorded by the Wearable Cardioverter Defibrillator
Acronym: ACAB
Status: Terminated | Type: Observational
Why Stopped: Unable to enroll suitable subjects
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90d0214
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Heart Failure Patients: Simultaneous recordings of cardiac acoustic biomarkers (CABs) by the Wearable Cardioverter Defibrillator and the AUDICOR AM
  Interventions: Device: Wearable Cardioverter Defibrillator

INTERVENTIONS:
Device: Wearable Cardioverter Defibrillator — Use of the Wearable Cardioverter Defibrillator and AUDICOR AM to evaluate accuracy of cardiac acoustic biomarker recordings.
  Other Names: AUDICOR AM

SUMMARY:
Evaluate data accuracy of cardiac acoustic biomarkers (CABs) recorded by the Wearable Cardioverter Defibrillator (WCD) as compared to the AUDICOR AM acoustic cardiography recorder.

DETAILED DESCRIPTION:
Single arm, prospective, non significant risk device study to evaluate data accuracy of cardiac acoustic biomarkers (CABs) recorded by the Wearable Cardioverter Defibrillator (WCD) compared with the CABs data simultaneously recorded by an acoustic cardiography recorder, the AUDICOR AM device.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* heart failure or a history of heart failure
* ischemic or non-ischemic cardiomyopathy
* ejection Fraction less than or equal to 40% as measured within the last 6 months

Exclusion Criteria:

* implanted left ventricular assist device
* pacemaker dependency
* currently hospitalized
* atrial fibrillation on their last ECG or having an irregularly irregular pulse

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary Care, Heart Failure, and Cardiology
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
CABs comparison | 2 hours
  Simultaneous CABs recordings from the AUDICOR and WCD devices will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Mike Osz, Study Director — Director, Clinical Operations, ZOLL
Locations (1):
- MAYO Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No